CLINICAL TRIAL: NCT05844111
Title: A Phase 1 Study To Investigate The Absorption, Metabolism, and Excretion of [14C]-BGB-11417 Following Single Oral Dose Administration in Healthy Male Subjects
Brief Title: A Study to Investigate the Absorption, Metabolism and Excretion of [14C]-BGB-11417
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BGB-11417-106
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C] radiolabeled BGB-11417 (Experimental): Participants will receive a single dose of [14C]-BGB-11417
  Interventions: Drug: [14C]-BGB-11417

INTERVENTIONS:
Drug: [14C]-BGB-11417 — A single oral dose of liquid formulation
  Other Names: Sonrotoclax

SUMMARY:
The main objective of this study is to determine the mass balance, routes of elimination, and pharmacokinetics of [14C]-BGB-11417 in healthy male participants along with determining the concentrations of radioactivity in plasma, fecal and urinary elimination of total radioactivity.

ELIGIBILITY:
Inclusion Criteria:

* The participant is judged by the investigator to be in good general health, as determined by no clinically significant findings from medical history, clinical laboratory assessments, vital sign measurements, 12-Lead electrocardiogram (ECG), and physical examination at screening and check-in
* The participant has a body mass index from 18.0 to 35.0 kilograms per square meter (kg/m^2), inclusive, at screening
* The participant has normal hepatic function (Note: Participants with Gilbert's syndrome should not be included)
* Participants must be willing to follow contraceptive practices, as applicable, from check-in until 90 days following study drug administration
* Participants must be willing to refrain from donating sperm from check-in until 90 days following study drug administration

Exclusion Criteria: -

* The participant has an absolute B-lymphocyte count of <200 cells/μL
* The participant has a medical history of any issues affecting swallowing, absorption, or metabolism, as judged by the investigator
* The participant has a medical history of any problems affecting venous access or bowel/bladder function
* The participant has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) types 1 or 2 antibodies at screening
* The participant is a smoker or has used nicotine or nicotine-containing products within 6 months before the first dose of study drug
* The subject has creatinine clearance of <90 mL/min, calculated with the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
* The participant has used any prescription or over-the-counter medications (except acetaminophen [up to 2 grams per day]), including herbal or nutritional supplements, within 14 days before the first dose of study drug
* The participant received any treatment with a moderate CYP3A4 inhibitor or strong CYP3A4 inducer within 14 days (or 5 half-lives, whichever is longer) before the first dose of study drug or during the study
* The participant has consumed grapefruit or grapefruit juice, Seville orange or Seville-orange-containing products (eg, marmalade), or caffeine- or xanthine-containing products within 48 hours before the first dose of study drug or during the study
* The participant has a history of alcohol abuse or drug addiction or psychiatric disorders including major depression disorder within the last year or excessive alcohol consumption (regular alcohol intake >21 units per week) (1 unit is equal to approximately one-half pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits
* The participant has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at screening or before the first dose of study drug.
* The participant is involved in strenuous activity or contact sports within 24 hours before the first dose of study drug or during the study

Note: Other inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-06-18 (Actual)

PRIMARY OUTCOMES:
Area under the concentration curve (AUC) from time 0 to the last quantifiable concentration (AUC0-t) of BGB-11417 | From 0 to 168 hours after study drug administration
Maximum concentration (Cmax) of BGB-11417 in Plasma | From 0 to 168 hours after study drug administration
Time to Cmax (Tmax) of BGB-11417 in Plasma | From 0 to 168 hours after study drug administration
Amount of BGB-11417-106 excreted (Ae) and Cumulative amount of BGB-11417-106 (Cum Ae) excreted in urine and feces | From 0 to 168 hours after study drug administration
Percentage (%Fe) and cumulative percentage (Cum %Fe) of BGB-11417 or radioactive dose excreted in urine and feces | From 0 to 168 hours after study drug administration

SECONDARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From the day of screening until end of study (approximately 1 month)

CONTACTS AND LOCATIONS:
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States